CLINICAL TRIAL: NCT01337375
Title: Pharmacokinetics and Pharmacodynamics of Intravenous Administration of Pegylated Interferon-2a in Patients With Chronic Hepatitis C and Previous Non-response to Standard Combination Therapy With Pegylated Interferon and Ribavirin (Intervention Study)
Brief Title: A Study of the Pharmacokinetics And Pharmacodynamics of Intravenously Administered Pegasys (Peginterferon Alfa-2a) in Patients With Chronic Hepatitis C And Previous Non-Response to Pegylated Interferon And Ribavirin Combination Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ML22936
Record Dates: First submitted 2011-03-29; First posted 2011-04-18 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a

ARMS (2):
- A/B (Experimental)
  Interventions: Drug: peginterferon alfa 2a [Pegasys]; Drug: peginterferon alfa-2a [Pegasys]
- C/D (Experimental)
  Interventions: Drug: peginterferon alfa-2a [Pegasys]

INTERVENTIONS:
Drug: peginterferon alfa 2a [Pegasys] — sc weekly
  Arms: A/B
Drug: peginterferon alfa-2a [Pegasys] — iv weekly
  Arms: A/B
Drug: peginterferon alfa-2a [Pegasys] — sc twice weekly
  Arms: C/D
Drug: peginterferon alfa-2a [Pegasys] — iv twice weekly
  Arms: C/D

SUMMARY:
In this randomized, cross-over, open label study the correlation of Pegasys (peginterferon alfa-2a) pharmacokinetics after intravenous (iv) and subcutaneous (sc) administration with viral load and viral kinetics will be investigated in patients with chronic hepatitis C genotype 1 who were non-responders to previous standard combination therapy with pegylated interferon and ribavirin. Patients will be randomized to receive either weekly or twice weekly Pegasys iv or sc for 2 weeks, crossing over to the other mode of administration after a washout period of 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult caucasian patients, 18 - 70 years of age
* Hepatitis C, genotype 1
* Non-responder to previous anti-HCV therapy with peginterferon alfa and ribavirin
* Compensated liver disease (Child-Pugh class A) for >/= 24 months before baseline
* Positive for anti-HCV for > 6 months, with detectable serum HCV-RNA

Exclusion Criteria:

* Treatment-naïve or responder to previous therapy
* HCV infection other than genotype 1
* Positive for Hepatitis A, Hepatitis B or HIV infection at screening
* Chronic Hepatitis of other than HCV origin
* Decompensated liver disease (Child-Pugh class B or C)
* Therapy with systemic antiviral, antineoplastic or immunomodulatory agents in the 6 months prior to study
* Clinically relevant retina disorder
* Pregnant or lactating women and male partners of pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
HCV RNA levels (IU/ml, COBAS TaqMan HCV Test) in correlation with area under the plasma concentration-time curve (AUC) after sc and iv administration | 11 months

SECONDARY OUTCOMES:
Evaluation of predictors of response to i.v. treatment | 11 months
Effect of waist to hip ratio on pharmacokinetics | 11 months
Effect of waist to hip ratio on viral response | 11 months
Incidence of adverse events | 11 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- Germany (5):
  - Berlin
  - Frankfurt am Main
  - Hamburg
  - Hanover
  - Leipzig